CLINICAL TRIAL: NCT01132170
Title: An Open Label, Balanced, Randomized, 2-treatment, 2-period, 2-sequence, Single Dose, Crossover, Bioequivalence Study of Divalproex Sodium DR 500 mg Tablets and Depakote® DR 500 mg Under Fasting Conditions.
Brief Title: Bioequivalency Study of Divalproex Sodium DR Tablets, 500 mg of Dr.Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Indu Bhushan / Senior Director R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-623/06-00
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Divalproex Sodium
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Divalproex Sodium DR Tablets 500 mg (Experimental): Divalproex Sodium DR Tablets 500 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Divalproex Sodium
- Depakote DR 500 mg Tablets (Active Comparator): Depakote DR 500 mg Tablets of Abbott Laboratories PR Ltd.,
  Interventions: Drug: Divalproex Sodium

INTERVENTIONS:
Drug: Divalproex Sodium — Divalproex Sodium DR Tablets 500 mg
  Other Names: Depakote DR 500 mg Tablets

SUMMARY:
The purpose of this study is to assess the bioavailability of Divalproex Sodium DR Tablets 500 mg versus Depakote DR 500 mg tablets with a washout period of 10 days in healthy subjects.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, bioequivalence study of Divalproex sodium DR 500 mg tablets of Dr.Reddy's Laboratories Limited, Generics, India comparing with that of Depakote® DR (containing Divalproex sodium) 500 mg tablets of Abbott Laboratories PR Ltd., Barceloneta, PR, in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

* Subjects who will provide written informed consent.
* Subjects must be healthy, adult, human beings within 18-45 years of age (both inclusive)weighing at least 50 kg.
* Having a Body Mass Index (BMI) between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m2
* Subjects must be of normal health as determined by medical history and physical examination performed within 21 days prior to the commencement of the study.
* Subjects whose screening laboratory values are within normal limits or considered by the physician/investigator to be of no clinical significance.
* Availability of the subject for the entire study period and willingness to adhere to the protocol requirements as evidenced by written informed consent.

Exclusion Criteria:

The subjects will be excluded based on the following criteria during screening and during the study

* Subjects incapable of understanding the informed consent.
* Subjects who have:

  * Systolic blood pressure less than 90 mm of Hg and more than 140 mm of Hg
  * Diastolic blood pressure less than 60 mm of Hg and more than 94 mm of Hg. Minor deviations (2-4 mm of Hg) at check-in may be acceptable at the discretion of the physician/investigator.
  * Pulse rate below 50/min and above 100/min.
* History of hypersensitivity or idiosyncratic reaction to Divalproex sodium or any other related drugs.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
* Consumption of grapefruit for the past ten days prior to the dosing day until the completion of the study.
* Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking from 48 hours before dosing and during sampling period
* Subjects who have taken over the counter or prescribed medications and enzyme modifying or any systemic medication for during the last 7 and 30 days respectively before dosing.
* Subjects who have participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.
* Subjects with clinically significant abnormalities (such as Laboratory Findings, ECG, X-Ray,Drugs of abuse, Alcohol etc.,) and/or with significant diseases (such as HIV, HCV, Syphilis,Hepatitis B etc.,).
* Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohanlal Siva Prasad Sayana, Principal Investigator — Bioserve Clinical Research Pvt. Ltd.,
Locations (1):
- Bioserve Clinical Research Pvt. Ltd.,, Hyderabad, Andhra Pradesh, India